CLINICAL TRIAL: NCT04515264
Title: The Association Between Human Milk Oligosaccharides (HMOs) Profiles and Growth Indicators of Infants Aged 0-4 Months. a Longitudinal Study
Brief Title: Human Milk Oligosaccharides (HMOs) Profiles and Growth Indicators of Infants Aged 0-4 Months
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Collaborators: Wyeth nutrition indonesia (Unknown)
Responsible Party: Principal Investigator, Verawati Sudarma, Principal Investigator, Indonesia University
Other Study IDs: HMOs Indonesia 1
Record Dates: First submitted 2020-08-13; First posted 2020-08-17 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Growth; Stunting, Nutritional
Keywords: human milk oligosaccharides
MeSH Terms: conditions — Growth Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The breastfeeding rates globally in Indonesia generally remain low with only 40% or less infants aged 6 months are exclusively breastfed. Available national data in 2018 showed the proportion of wasted in children under 5 years old was 6.7%, while 3.5% children were severely wasted. This data showed improvement compared data in 2007 and 2013. While proportion children under 2 years old with stunted and severly stunted was 29.9%. As the third most abundant group of compounds in human milk, after lactose (70 g/L) and lipids (40 g/L), human milk oligosaccharides (HMOs) never been study in Indonesia. HMOs amount and diversity influenced by non modifiable and modifiable factors. The maternal phenotypes, the α-1-2-fucosyltransferase (FUT-2) gene and the α-1-3-4-fucosyltransferase (FUT-3) gene divided the mother into secretor (Se+) and non secretor (Se-) and Le+ or Le-). Studies showed the breastfed infants of non secretor mothers secrete lower HMOs than secretor mothers. By many functions in HMOs such as prebiotic, anti infection, modulate immunity, it is thought that HMOs can influence infant growth. The hypothesis of this study is to show the associations between maternal factors (secretor gene status/FUT-2 gene, lewis gene status/FUT-3 gene, gestational age and gestational weight gain) with HMOs profiles and growth indicators of infants aged 0-4 months.

DETAILED DESCRIPTION:
This study is a prospective longitudinal study to analyze the association between HMOs profiles and growth indicators of infants age 0-4 months. In this longitudinal study, the human milk, anthropometry assessment and questionnaires will be collect in the 0, 2, 4 month of age. Gestational age and birth weight will be obtain from the medical status upon enrollment.

The study will be conduct in Government & Private Hospital in Jakarta between Juli - December 2020. Based on sample size calculation, the total minimal samples are 120 samples. Subjects recruitment will be based on nonprobabilistic consecutive sampling to post partum inpatient mothers in Government & Private Hospital in Jakarta between Juli - December 2020.

Study forms consist of study information, informed consent, screening form, baseline data, follow up form and laboratory result form. The tools requirements are among others Seca 728 electronic infant scale, Anthropometry Plus (AnthroPlus) Software, World Health Organization (WHO) growth velocity chart, Questionnaires, Thermometer, 15 mL polypropylene tube, Disposable gloves and vacuum bag with dry ice. The specimens obtain for this study are 15 mL venous blood for genotyping and 10 mL breast milk (0, 2, 4 month).

After obtaining clearance from Ethical Committee of the Faculty of Medicine University of Indonesia, the post partum mothers will be presented with Form A (study information form). Patients will be informed about the aim, benefits and procedures of the study. If patients agree, she will have to sign the informed consent (Form B).

Study phases consists of

1. screening : description of the aims, benefits and procedures of the study, filling the informed consent, screening based on inclusion and exclusion criteria.
2. Data collection :

   * Interview. Interview will be done to fill information in Form C and D.
   * Subjects selected during the screening visit will follow a 4 month study. Primary and secondary outcomes will be measured at 0, 2, 4 months (visit 1-2-3).
3. Data analysis :

   1. All data will be edited, coded and entry to the computer. The Statistical Package for the Social Sciences (SPSS) for windows version 20.0 will be use for data analyzing.
   2. Univariate analysis will be conduct to know the distribution of each variables. Test of normality of the data will be perform with Kolmogorov-Smirnov test at the significance level p>0.05 as normally distributed data. The continuous data will be present as mean ± standard deviation and for categorical data in n (%) for normally distributed data and geometric mean ± standard deviation forn non-normally distributed data.
   3. For bivariate analysis, Pearson correlation test will be performed if the data is normally distributed or Spearman Rank test if the data is non-normally distributed. Reference for rho value show in Table 3.3.
   4. Multivariate analysis will be conduct by linear regression model.

ELIGIBILITY:
Inclusion Criteria:

Mother :

* Age of 18-45 year at the time of delivery
* Willing to breastfed at least up to 4 month
* Singleton birth

Exclusion Criteria:

* Mother :

  * Type 1 or 2 diabetes before or during pregnancy
  * Presenting conditions that contraindicate breastfeeding
  * Smoking
* Infant :

  * Congenital illness or malformation that could affect growth
  * Infants received water or any other food besides breast milk

Ages: 2 Weeks to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Target population of this study are post partum inpatient mothers in Government & Private Hospital in Jakarta between July - Agustus 2020.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-04-22 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Weight for Age Z score (WAZ) | Change from baseline WAZ at 2 months.
  weight-for-age z score WHO growth chart. Comparing the weight of infant with age based on WHO growth chart.
Weight for Age Z score (WAZ) | Change from baseline WAZ at 4 months.
  weight-for-age z score WHO growth chart. Comparing the weight of infant with age based on WHO growth chart.
Weight for Length Z score (WLZ) | Change from baseline WLZ at 2 months.
  weight-for-length z score WHO growth chart. Comparing the weight of infant with length based on WHO growth chart.
Weight for Length Z score (WLZ) | Change from baseline WLZ at 4 months.
  weight-for-length z score WHO growth chart. Comparing the weight of infant with length based on WHO growth chart.
Weight velocity | Change from baseline weight velocity at 2 months.
  Comparing the infant weight gain with weight velocity chart from WHO
Weight velocity | Change from baseline weight velocity at 4 months.
  Comparing the infant weight gain with weight velocity chart from WHO

CONTACTS AND LOCATIONS:
Overall Officials: Verawati Sudarma, Master, Principal Investigator — Indonesia University
Locations (1):
- Universitas Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No
The Individual participant data (IPD) will be shared based on request